CLINICAL TRIAL: NCT00292942
Title: A Phase 1 Double-Blind, Placebo-Controlled, Randomized Multiple Dose Escalation Study to Evaluate the Safety, Tolerance, and Pharmacokinetics/Pharmacodynamics of a New GMP Formulation of Intravenous Artesunate if Healthy Subjects
Brief Title: Study of the Safety of Intravenous Artesunate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WRAIR 1142; USUHS G183SP (Other); A-13419 (Other: IRB)
Record Dates: First submitted 2006-02-14; First posted 2006-02-16 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-02

CONDITIONS: Malaria; Malaria, Cerebral
Keywords: artesunate; artemisinin; falciparum
MeSH Terms: conditions — Malaria; Malaria, Cerebral | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 2 mg/kg Intravenous Artesunate (Experimental): 2 mg/kg of Intravenous artesunate
  Interventions: Drug: Intravenous Artesunate
- 4 mg/kg Intravenous Artesunate (Experimental): 4 mg/kg of Intravenous artesunate
  Interventions: Drug: Intravenous Artesunate
- 8 mg/kg Intravenous Artesunate (Experimental): 8 mg/kg of Intravenous artesunate
  Interventions: Drug: Intravenous Artesunate
- Placebo (Placebo Comparator): Mannitol (200 mg/vial) diluted in phosphate buffer and delivered in an equivalent volume by subject's weight as artesunate.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravenous Artesunate — Three doses of Intravenous Artesunate drug at 2, 4, or 8 mg/kg in diluent Phosphate Buffer (0.3 M, pH 8.1)
  Other Names: IV AS
  Arms: 2 mg/kg Intravenous Artesunate; 4 mg/kg Intravenous Artesunate; 8 mg/kg Intravenous Artesunate
Drug: Placebo — Mannitol (200 mg/vial) diluted in Phosphate Buffer and given IV in equivalent volume by subject's weight.
  Other Names: Mannitol
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish the safety, tolerability, and pharmacokinetics of a multiple dose of the antimalarial drug artesunate.

DETAILED DESCRIPTION:
This study was a Phase 1b, randomized, double-blind, placebo-controlled trial using multiple ascending doses of intravenous artensunate (AS) to determine it's safety, tolerability, and PK in healthy subjects. Subjects were screened within 21 days of dosing. At the screening visit, subject underwent baseline assessments: vital signs were recorded; a physical examination, urinalysis, urine drug screen, and urine pregnancy test were performed; a complete blood cell count (CBC) with differential and indices, reticulocyte count, coagulation markers, and blood chemistry assessments were performed and medical and medication history was collected. Eligible subjects were scheduled for a 6-hour pre-dose electrocardiogram (ECG) and vital sign assessment with measurements taken at approx. the same times as Day 1 (dosing day). On Day 0, subjects were admitted to the clinical pharmacology unit to begin the inpatient phase of the study. Subjects had a brief physical examination and all procedures for the inpatient stay were reviewed. On Day 1, pre-dose vital signs and ECG were performed. Subjects then received study drug or placebo by IV bolus infusion. Subjects were closely monitored by evaluating hemodynamic measurements, periodic ECGs, and assessment of spontaneously reported AEs. Blood was drawn for blood count and chemistry analysis 6h and 24h after each dose. PK blood samples were drawn pre-dose and approx. 5min, 20min, 40min, 1h, 2h, 4h, 6h, and 24h after each dose. On Days 2 and 3 subjects received their second and third doses, respectively, of study drug or placebo with the same monitoring and laboratory measurements as for the first dose. Subjects were discharged 24 hours after the 3rd dose of drug or placebo and were followed as outpatients on Days 7, 10, and 15.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and non-pregnant, non-lactating females
* Have a normal ECG that may include benign PAC's and PVC's, 1st degree AV block, 2nd degree AV block, Wenckebach
* Have a normal blood pressure (BP) and heart rate (HR). These will be measured after resting supine for about 3 minutes. Normal BP is defined as less than 140 mm Hg systolic and less than 90 mm Hg diastolic. Normal baseline HR is 50 to 90 bpm without symptoms.
* Body mass index between 18 and 29 kg/m**2 or, if out of range, not clinically significant (within 15% of their ideal body weight).
* Be able to verbalize understanding of the consent form, provide written informed consent and verbalize willingness to complete study procedures
* Have a physical examination that demonstrates no clinically significant contraindication for participating in the study. This would include documentation of any abnormal movements suggesting neurological pathology and ECG tracings to document an abnormalities in cardiac conduction
* If female, have a negative serum pregnancy test at screening and urine pregnancy test on pre-admission and admission, or be postmenopausal, or have had a hysterectomy, or have been sterilized, AND, if still able to bear children, agree to practice effective contraception for the duration of the study and for a period of 12 weeks after stopping study drug.
* Active duty participants must be on leave during the inpatient phase of the study.

Exclusion Criteria:

* Have received any investigational drug or vaccine in the period 0 to 16 weeks before entry to the study.
* Have been on a liquid protein diet in the last year
* Have any clinically important physical findings, laboratory abnormalities, or histories of Rx or OTC drug use that may, in the judgement of a study investigator, impact study interpretation or affect subject safety
* Have used any prescription drugs within 14 days prior to admission or most non-prescription drugs including herbals or dietary supplements within 7 days prior to admission (at the investigator's discretion).
* Existence of any surgical or medical condition that, in the judgement of the clinical investigator, might interfere with the distribution, metabolism or excretion of the drug
* Presence of history of drug allergy requiring treatment. Hay fever is allowed unless it is active or has required treatment within the previous 2 months
* Donation or loss of greater than 400 ml of blood in the period 0 to 12 weeks before entry to the study.
* Serious adverse reaction or hypersensitivity to any drug, particularly artemisinin derivatives
* CAGE (screening test for alcoholism) postitive (2 out of 4 criteria) or has a history of recent alcohol abuse
* Use of illicit drugs
* Family history (in 1st degree relatives) of sudden cardiac death or prolonged QT/QTc syndrome
* History of seizure (excluding febrile seizures in childhood), episodes of unexplained syncope, or trouble with balance, undiagnosed hearing deficits, and other neurological disorder
* History of severe psychiatric disorder or hospitalization for severe psychiatric disorder
* Current job or personal habit of reversed sleep-wake cycle
* History of cardiac disease to include cardiomyopathy, valvular disease, arrhythmia, ischemia, or enlarged heart
* Presence of hepatitis B surface antigen (Hbs-Ag), hepatitis C antibody (antiHCV) or HIV type 1 at screening
* A finding or history of hematuria (excluding menses-related hematuria) during subject screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-06-12 (Actual); Primary Completion 2007-01-17 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Weina, MD, PhD, Study Director — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Uniformed Services University of the HEalth Sciences, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
WRAIR

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 47 subjects were screened over the 3 dose escalation cohorts of the study. Twenty-six subjects were enrolled and received IV AS at the USUHS, Clinical Pharmacology Unit (CPU), Bethesda, MD
Period: Overall Study
Arm/Group | Placebo | 2 mg/kg Intravenous Artesunate | 4 mg/kg Intravenous Artesunate | 8 mg/kg Intravenous Artesunate
Started | 6 | 6 | 7 | 7
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2 mg/kg Intravenous Artesunate | 4 mg/kg Intravenous Artesunate | 8 mg/kg Intravenous Artesunate | Total
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (10.41) | 43.2 (12.02) | 35.3 (9.96) | 35.0 (11.86) | 37.2 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 2
  Male | 5 | 6 | 6 | 7 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 4 | 3 | 3 | 12
  Black or African American | 4 | 0 | 2 | 3 | 9
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0
  Subjects with >1 race | 0 | 2 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 7 | 7 | 26
Height (cm) [Mean (Standard Deviation); unit: cm] | 173.68 (7.598) | 172.97 (3.634) | 173.14 (12.472) | 175.34 (2.519) | 173.82 (7.348)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 80.33 (8.390) | 76.53 (11.114) | 81.03 (12.681) | 77.80 (5.912) | 78.96 (9.445)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.68 (2.917) | 25.50 (2.828) | 26.89 (2.270) | 25.30 (1.628) | 26.09 (2.386)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With AEs
Description: The general strategy of the safety analysis was to examine the clinical tolerability and laboratory safety parameter data and determine if there were any trends amongst the dose levels concerning all AEs and drug related AEs.
Time Frame: up to 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 2 mg/kg Intravenous Artesunate | 4 mg/kg Intravenous Artesunate | 8 mg/kg Intravenous Artesunate
Number analyzed (Participants) | 6 | 6 | 7 | 7
Participants
  All AEs: No AEs | 0 | 0 | 2 | 0
  All AEs: Subjects with 1 AE | 3 | 3 | 0 | 2
  All AEs: Subjects with 2 AEs | 3 | 0 | 1 | 2
  All AEs: Subjects with ≥3 AEs | 0 | 3 | 4 | 3
  Drug Related AEs: No AEs | 2 | 0 | 2 | 1
  Drug Related AEs: Subjects with 1 AE | 2 | 3 | 1 | 2
  Drug Related AEs: Subjects with 2 AEs | 2 | 1 | 1 | 2
  Drug Related AEs: Subjects with ≥3 AEs | 0 | 2 | 3 | 2

2. Primary Outcome: Number of Participants With AEs Occurring in Greater Frequency in the 2.0 mg/kg IV AS Group Then in the Placebo Group to Access Safety and Tolerability of AS
Description: Comparison of number of participants with AEs reported for the placebo control and those treated with the 2.0 mg/kg of IV AS to access safety and tolerability
Time Frame: up to 21 days
Population: As the intended, compassionate use dose of Intravenous Artesunate will be 2.4 mg/kg for the treatment of individuals with severe malaria, a comparison was performed between the frequency of AEs reported for the placebo control subjects and those treated with the 2.0 mg/kg dose of Intravenous Artesunate.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 2 mg/kg Intravenous Artesunate
Number analyzed (Participants) | 6 | 6
Participants
  Dysguesia | 1 | 4
  Dizziness | 0 | 1
  Headache | 1 | 3
  Parethesia | 0 | 1
  Parosmia | 0 | 1
  Erythema | 0 | 1
  Pruritus Generalized | 0 | 1
  Tenderness | 0 | 1
  Venipuncture Site Inflammation | 0 | 1
  Eye Pain | 0 | 1
  Back Pain | 0 | 1
  Muscle Strain | 0 | 1

3. Secondary Outcome: Cardiovascular Responses: Number of Participants With Changes in Blood Pressure and Heart Rate After Infusion
Description: Cardiovascular Responses: Number of participants with changes in blood pressure and heart rate after infusion to determine change from baseline
Time Frame: screening, on Day -1, on Days 1, 2, and 3, and at each follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 2 mg/kg Intravenous Artesunate | 4 mg/kg Intravenous Artesunate | 8 mg/kg Intravenous Artesunate
Number analyzed (Participants) | 6 | 6 | 7 | 7
Participants
  Systolic BP change of at least 20mmHg: Increase | 1 | 1 | 1 | 1
  Systolic BP change of at least 20mmHg: Decrease | 0 | 0 | 0 | 0
  Systolic BP change of at least 20mmHg: No significant change | 5 | 5 | 6 | 6
  Heart Rate change of at least 15bpm: Increase | 4 | 4 | 6 | 3
  Heart Rate change of at least 15bpm: Decrease | 0 | 0 | 0 | 0
  Heart Rate change of at least 15bpm: No significant change | 2 | 2 | 1 | 4

4. Secondary Outcome: Range of Pharmacokinetic Parameters for Artesunic Acid After Single 2.0, 4.0 and 8.0 mg/kg Dose of Artesunate Daily for 3 Days (ng*hr/mL)
Description: For artesunic acid, AUC0-last was determine for each dose; as well as the total area under the curve (AUClastTOTAL), calculated as the sum of AUClast for each of the doses (ng*hr/mL)
Time Frame: Pre-dose, 5, 20, 40 minutes after infusion and 1, 2, 4, 8, 24 and 72 hours after infusion
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | 2 mg/kg Intravenous Artesunate | 4 mg/kg Intravenous Artesunate | 8 mg/kg Intravenous Artesunate
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL
  AUC24 1 (ng.hr/mL) | 1368 (912) | 2325 (721) | 5766 (2121)
  AUC24 2 (ng.hr/mL) | 978 (648) | 1746 (247) | 5272 (2089)
  AUC24 3 (ng.hr/mL) | 935 (301) | 1880 (795) | 4379 (2361)
  AUC last 1 (ng.hr/mL) | 1162 (656) | 2421 (755) | 4631 (2402)
  AUC last 2 (ng.hr/mL) | 932 (524) | 1636 (342) | 5728 (1980)
  AUC last 3 (ng.hr/mL) | 933 (239) | 1627 (957) | 4374 (2362)
  AUC last TOTAL (ng.hr/mL) | 3027 (1158) | 5683 (550) | 14733 (5846)

5. Secondary Outcome: Range of Pharmacokinetic Parameters for Artesunic Acid After Single 2.0, 4.0 and 8.0 mg/kg Dose of Artesunate Daily for 3 Days (ng/mL)
Description: For the predicted concentration at the time of dose administration (C0) was determine for each dose (ng/mL)
Time Frame: Pre-dose, 5, 20, 40 minutes after infusion and 1, 2, 4, 8, 24 and 72 hours after infusion
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 2 mg/kg Intravenous Artesunate | 4 mg/kg Intravenous Artesunate | 8 mg/kg Intravenous Artesunate
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  C0 1 | 14840 (10902) | 29056 (12850) | 53503 (33017)
  C0 2 | 11992 (8311) | 17265 (3590) | 66380 (32973)
  C0 3 | 10408 (1851) | 23417 (10200) | 54674 (43261)

6. Secondary Outcome: Range of Pharmacokinetic Parameters for Dihydroartemisinin (DHA) After Single 2.0, 4.0 and 8.0 mg/kg Dose of Artesunate Daily for 3 Days (ng*hr/mL)
Description: For DHA, AUC24, and AUClast were calculated for each dose, as well as the total area under the curve extrapolated to infinite time (AUC∞TOTAL), calculated as the sum of AUC24 for each dose +C24/λz.
Time Frame: Pre-dose, 5, 20, 40 minutes after infution and 1, 2, 4, 8, 24 and 72 hours after infusion
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | 2 mg/kg Intravenous Artesunate | 4 mg/kg Intravenous Artesunate | 8 mg/kg Intravenous Artesunate
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL
  AUC24 1 | 1982 (377) | 4122 (809) | 8992 (3355)
  AUC24 2 | 1865 (512) | 3509 (970) | 8122 (2750)
  AUC24 3 | 2204 (524) | 3748 (646) | 8571 (2817)
  AUC last 1 | 1954 (367) | 4065 (771) | 8842 (3265)
  AUC last 2 | 1847 (516) | 3394 (974) | 8011 (2780)
  AUC last 3 | 2171 (519) | 3701 (647) | 8405 (2715)
  AUC oo TOTAL | 6051 (1074) | 11379 (2128) | 25685 (8715)

7. Secondary Outcome: Cmax Assessment After Single 2.0, 4.0 and 8.0 mg/kg Dose of Artesunate Daily for 3 Days (ng/mL)
Description: Cmax was calculated after single 2.0, 4.0 and 8.0 mg/kg dose of Artesunate daily for 3 days (ng/mL)
Time Frame: Pre-dose, 5, 20, 40 minutes after infution and 1, 2, 4, 8, 24 and 72 hours after infusion
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 2 mg/kg Intravenous Artesunate | 4 mg/kg Intravenous Artesunate | 8 mg/kg Intravenous Artesunate
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Cmax 1 | 1735 (547) | 3015 (882) | 6057 (2456)
  Cmax 2 | 1710 (715) | 2923 (1050) | 5943 (2110)
  Cmax 3 | 2358 (634) | 2933 (810) | 5762 (3426)

8. Secondary Outcome: Tmax Assessment After Single 2.0, 4.0 and 8.0 mg/kg Dose of Artesunate Daily for 3 Days (hr)
Description: Tmax was calculated after single 2.0, 4.0 and 8.0 mg/kg dose of Artesunate daily for 3 days (hr)
Time Frame: Pre-dose, 5, 20, 40 minutes after infution and 1, 2, 4, 8, 24 and 72 hours after infusion
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | 2 mg/kg Intravenous Artesunate | 4 mg/kg Intravenous Artesunate | 8 mg/kg Intravenous Artesunate
Number analyzed (Participants) | 6 | 6 | 6
hr
  Tmax 1 (hr) | 0.244 (0.132) | 0.208 (0.137) | 0.208 (0.137)
  Tmax 2 (hr) | 0.167 (0.129) | 0.208 (0.137) | 0.181 (0.238)
  Tmax 3 (hr) | 0.122 (0.104) | 0.292 (0.102) | 0.250 (0.129)

ADVERSE EVENTS:
Time Frame: up to 21 days
Arm/Group | Placebo | 2 mg/kg Intravenous Artesunate | 4 mg/kg Intravenous Artesunate | 8 mg/kg Intravenous Artesunate
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/7 | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | 2 mg/kg Intravenous Artesunate (N=6) | 4 mg/kg Intravenous Artesunate (N=7) | 8 mg/kg Intravenous Artesunate (N=7)
Dysgeusia (Nervous system disorders) | 1 (1) | 4 (4) | 6 (6) | 6 (6)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venipuncture site (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No